CLINICAL TRIAL: NCT01982695
Title: Compare Efficacy of the Angiotensin Converting Enzyme Inhibitor (ACEi) Lisinopril With Angiotensin II Receptor Antagonist Losartan (ARB) for the Cardiomyopathy of Duchenne Muscular Dystrophy
Brief Title: Cardiomyopathy in DMD: Lisinopril vs. Losartan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Boston Children's Hospital (Other); University of California, Davis (Other); University of Kansas Medical Center (Other); University of Minnesota (Other); St. Louis Children's Hospital (Other)
Responsible Party: Principal Investigator, Jerry R. Mendell, Director, Center for Gene Therapy, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB12-00149
Record Dates: First submitted 2013-10-29; First posted 2013-11-13 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-01

CONDITIONS: Duchenne Muscular Dystrophy (DMD); Cardiomyopathy
Keywords: Duchenne muscular Dystrophy (DMD); Cardiomyopathy; Losartan; Lisinopril
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Cardiomyopathies | interventions — Losartan; Lisinopril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lisinopril (Active Comparator)
  Interventions: Drug: Lisinopril
- Losartan (Active Comparator)
  Interventions: Drug: Losartan

INTERVENTIONS:
Drug: Losartan
  Arms: Losartan
Drug: Lisinopril
  Arms: Lisinopril

SUMMARY:
This trial is a double-blind randomized clinical trial of lisinopril versus losartan for the treatment of cardiomyopathy in Duchenne Muscular Dystrophy (DMD). Both drugs are known to be effective for the treatment of dilated cardiomyopathy. ACEi have been reported to delay the onset and progression of left ventricle dysfunction in children with DMD. Multiple studies show therapeutic efficacy of losartan in animals with cardiomyopathy related to muscular dystrophy and in patients with cardiomyopathy from diverse causes. ARBs are often reserved for patients in whom heart failure is not adequately treated or where side effects preclude the use of an ACEi. However, in DMD, losartan might be a better choice as a first line drug because of studies demonstrating a potential benefit for skeletal muscle in the mdx mouse. Considering that both skeletal and cardiac muscles are major contributors of the disability of DMD, a drug that could improve both heart and skeletal muscles simultaneously would need consideration as the drug of choice for the cardiomyopathic DMD patient.

ELIGIBILITY:
Inclusion Criteria:

* Duchenne muscular dystrophy patients of all ages
* Null mutation of the dystrophin gene or muscle with <5% dystrophin
* Doppler echocardiogram with ejection fraction (EF) <55% within 30 days of enrollment
* Ability to cooperate for testing
* Glucocorticoid treatment acceptable including daily or weekend administration of prednisone or deflazacort

Exclusion Criteria:

* Patients with EF 55% or greater
* Patients with EF <40% after washout
* Patients taking >5 mg lisinopril, or >25 mg losartan or >5 mg enalapril
* Skeletal deformities or pulmonary anatomical variants that preclude consistent measures of Doppler echocardiography

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-03; Primary Completion 2012-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California Davis, Davis, California
  - University of Kansas Medical Center, Kansas City, Kansas
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota, Saint Paul, Minnesota
  - St. Louis Children's Hospital, Saint Louise, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio

REFERENCES:
- [Background] Thrush PT, Allen HD, Viollet L, Mendell JR. Re-examination of the electrocardiogram in boys with Duchenne muscular dystrophy and correlation with its dilated cardiomyopathy. Am J Cardiol. 2009 Jan 15;103(2):262-5. doi: 10.1016/j.amjcard.2008.08.064. Epub 2008 Oct 30. PMID 19121448
- [Result] Viollet L, Thrush PT, Flanigan KM, Mendell JR, Allen HD. Effects of angiotensin-converting enzyme inhibitors and/or beta blockers on the cardiomyopathy in Duchenne muscular dystrophy. Am J Cardiol. 2012 Jul 1;110(1):98-102. doi: 10.1016/j.amjcard.2012.02.064. Epub 2012 Mar 29. PMID 22463839
- [Derived] Allen HD, Flanigan KM, Thrush PT, Dvorchik I, Yin H, Canter C, Connolly AM, Parrish M, McDonald CM, Braunlin E, Colan SD, Day J, Darras B, Mendell JR. A randomized, double-blind trial of lisinopril and losartan for the treatment of cardiomyopathy in duchenne muscular dystrophy. PLoS Curr. 2013 Dec 12;5:ecurrents.md.2cc69a1dae4be7dfe2bcb420024ea865. doi: 10.1371/currents.md.2cc69a1dae4be7dfe2bcb420024ea865. PMID 24459612
- See also: Center for Gene Therapy, The Research Institute at Nationwide Children's Hospital — http://www.nationwidechildrens.org/center-for-gene-therapy
- See also: The Muscular Dystrophy Association — http://mdausa.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Lisinopril: Approximately 0.07 mg/kg/day in oral capsules
- Losartan: Approximately 0.7 mg/kg/day in oral capsules
Period: Overall Study
Arm/Group | Lisinopril | Losartan
Started | 12 | 11
Completed | 12 | 10
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Lisinopril; Lospartan: Lisinopril
- Total: Total of all reporting groups
Arm/Group | Lisinopril | Lospartan | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Median (Full Range); unit: years] | 12.5 [10 to 21] | 15.5 [7 to 27] | 14 [7 to 27]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 11 | 23
Ejection Fraction [Mean (Standard Deviation); unit: percentage of blood leaving the heart] | 47.5 (6.25) | 47.7 (5.49) | 47.6 (5.77)

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Ejection Fraction as Measured by Echocardiogram
Description: Mean cardiac ejection fraction as measured by echocardiogram at 12 month study visit. Cardiac ejection fractions were measured using the biplane Simpson's rule using images obtained from the apical 4 chamber views of the heart.
Time Frame: 12 month visit
Population: All patients that received a 12 month echocardiogram evaluation
Measure: Mean (Standard Deviation); unit: percentage of blood leaving the heart
Groups:
- Losartan: Losartan
Arm/Group | Lisinopril | Losartan
Number analyzed (Participants) | 7 | 9
percentage of blood leaving the heart | 54.6 (5.19) | 55.2 (7.19)

ADVERSE EVENTS:
Arm/Group | Lisinopril | Losartan
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisinopril (N=12) | Losartan (N=10)
Allergic reaction to medication (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes